CLINICAL TRIAL: NCT04987060
Title: Intrastromal Fresh Human Corneal Lenticule Implantation Using Smile Surgery for Treatment of Irregular Corneal Astigmatism After Penetrating Keratoplasty (new Approach)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye Hospital Pristina Kosovo (Other)
Responsible Party: Principal Investigator, Dr. Faruk Semiz, Head of Ophthalmology Department, Eye Hospital Pristina Kosovo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EyeHPristina2
Record Dates: First submitted 2021-07-27; First posted 2021-08-03 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-02

CONDITIONS: Irregular Astigmatism

STUDY DESIGN:
Intervention Model Description: Irregular astigmatism group
Masking Description: irregullar astigmatism group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intrastromal Fresh Human Lenticule Implantation (Other): The aim of this study is to investigate the effect of intrastromal fresh corneal lenticule implantation using Smile module surgery after PK with primary objective to increase visual acuity by reducing irregular astigmatism according to high K values. The stromal pocket diameter was 8 mm, 2mm super incision, 140-µm cap thickness and fresh lenticular implantation is performed.
  Interventions: Device: Intrastromal Fresh Human Lenticule Implantation

INTERVENTIONS:
Device: Intrastromal Fresh Human Lenticule Implantation — The stromal pocket diameter was set 8.0 mm and cap thickness was set to 140 μm from corneal surface and a 2mm superior incision. Hinge position flap was set at 90°, angle 50° and width 4 mm, side cut angle 90°. The pocket was dissected using a blunt spatula washed with normal saline. The lenticule was held with lenticule forceps and gently inserted into the pocket through the 2 mm superior incision. Incision position changed according to the position of the highest K values.

SUMMARY:
The aim of the study is to present the effect of implanting intrastromal fresh corneal lenticule by SMILE surgery as a new method-approach to correct the corneal shape on purpose to reduce irregular astigmatism and increasing visual acuity after penetrating keratoplasty.

DETAILED DESCRIPTION:
Irregular astigmatism occurs when the curvature of the eye is pronounced in any direction, not just the center. The curve could be steeper towards the bottom than on top, or it could be any configuration in which the eye's surface area is uneven.

Irregular astigmatism usually can result from corneal degenerations(keratoconus,pellucid marginal degeneration,keratoglobus), corneal surgery or trauma.

Irregular astigmatism is still the main cause of decreased visual acuity after penetrating keratoplasty.

Our study present new therapeutic method and new technology to manage irregular astigmatism after PK. Knowing that the incidence of high and irregular astigmatism after PK is still a frequent complication and source of frustration for patients and corneal surgeons our study present an adequate surgical technique implanting intrastromal human corneal lenticule using SMILE for treatment of corneal irregular astigmatism after PK trying satisfy patients visual expectations.

ELIGIBILITY:
Inclusion Criteria:

* patients with irregular astigmatism
* low visual acuity

Exclusion Criteria:

* history of glaucoma
* retinal detachment
* history of ocular inflamation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Increase of visual acuity | 12 months
  Using intrastromal fresh corneal lenticule resulted in the increase of the visual acuity.

SECONDARY OUTCOMES:
Decrease of irregular astigmatism | 12 months
  In order to stabilize irregular astigmatism and reduce K-values, the intrastromal fresh corneal lenticule was implanted.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital Pristina, Pristina, Kosovo

IPD SHARING:
Plan to Share IPD: Undecided